CLINICAL TRIAL: NCT01847040
Title: Deployment Related Mild Traumatic Brain Injury (mTBI): Incidence, Natural History, and Predictors of Recovery in Soldiers Returning From OIF/OEF
Brief Title: Deployment Related Mild Traumatic Brain Injury (mTBI)
Status: Completed | Type: Observational
Sponsor: The Defense and Veterans Brain Injury Center (U.S. Federal Agency)
Collaborators: VISN 19 Mental Illness, Research, Education and Clinical Center (U.S. Federal Agency); Womack Army Medical Center (U.S. Federal Agency); USUHS Preventive Medicine and Biometrics (Unknown)
Responsible Party: Principal Investigator, Karen Schwab, Chief, Epidemiology and Research Support, The Defense and Veterans Brain Injury Center
Other Study IDs: W81XWH-08-2-0105
Record Dates: First submitted 2013-04-26; First posted 2013-05-06 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2013-05

CONDITIONS: Mild Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Epidemiology; Concussion; Outcomes; PTSD; Prospective; Longitudinal; Military; Symptoms; Validation; Screening; Mild Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion; Brain Injuries, Traumatic; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- TBI while Deployed: Active duty service members returning from Afghanistan or Iraq who were screened positive for Mild TBI
- No TBI while Deployed: Active duty service members returning from Afghanistan or Iraq who screened negative for mild TBI.

SUMMARY:
The study will provide evidence on the long term outcomes of mTBI in service members returning from Afghanistan and Iraq. In addition, the study will provide evidence on mTBI incidence, and symptom patterns. Self-reported assessments at baseline and follow-ups will be combined with data on health care utilization and military job performance. The work, symptoms, and family interaction outcomes of returning soldiers screening positive for mTBI, combined mTBI and PTSD, and soldier controls will be compared at 3 months, 6 months, and at one year. The assessments over time will permit descriptions of symptom changes for these populations. It is likely the study will find similar findings to those of previous civilian studies - that concussive symptoms often resolve within months of injury. However, some soldier subsets may have chronic problems. Determining the incidence and outcomes of individuals with mTBI will assist medical providers in determining the types of follow-ups needed by returning service members and suggest the development of additional treatment interventions. These results may also inform treatment of civilian populations with mTBI.

The three primary hypotheses are:

1. Concussive symptoms at the time of return from serving in Afghanistan and Iraq and symptoms persisting 3 months, 6 months, and 12 months after return will be associated with extent of exposure to combat, injury mechanism, associated injuries (co-occuring injuries), PTSD and other psychiatric co-morbidities, and number of deployment-related mTBIs.
2. Returning troops reporting concussive symptoms at the time of return from deployment will have more work related problems at each follow-up (including lower rates of return to duty, return to work, and poor quality of work).
3. The mTBI screening tool will be sensitive and specific to mTBI when compared to the criterion measure, which is a structured interview conducted by clinicians blinded to the screening results.

ELIGIBILITY:
Inclusion Criteria:

1. Must be returning from deployment in Iraq or Afghanistan
2. Must have been screened for mild TBI on the deployment related study screening tool
3. Must sign an informed consent/HIPAA authorization -

Exclusion Criteria:

1. Returning from deployment for medical reasons, that is, medically evacuated to the Continental US
2. Unable or unwilling to provide informed consent/HIPAA authorization -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cohort of soldiers returning to Fort Bragg and Fort Carson returning from deployment to Iraq and Afghanistan. National Guard and Army Reservists serving on Active Duty will also be included.
Sampling Method: Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2009-09; Primary Completion 2013-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Over time change in Concussive symptoms | Baseline; 3 months; 6 months; 12 months
  Concussive symptoms are measured with 3 instruments: Neurobehavioral Symptom Inventory; Patient Health Questionnaire; Headache Questionnaire.
Change in Work Related Issues | 3 months; 6 months; 12 months
  Measures of rates of return to duty; rates of return to work; and military job performance (for subjects remaining in military at follow-up).

SECONDARY OUTCOMES:
Automated Neuropsychological Assessment Metrics (ANAM) | Pre-deployment testing; and upon return from deployment
  The ANAM is a brief computerized cognitive assessment tool used for all individuals deploying to Afghanistan or Iraq; and administered after return from deployment.
Change in Social Interaction | Baseline; 3 months; 6 months; 12 months
  Quality and frequency of interactions with family, friends, and partners. Includes marital status, living arrangements, best friend, people can depend upon for help, comparative quality of relationships before deployment and currently, frequency of communication.
Alcohol and caffeine use | Baseline; 3 months; 6 months; 12 months
  Frequency of alcohol consumption, pre and post deployment consumption, receipt of help.
  Frequency of caffeine consumption, amount, consume with alcohol.
Health Utilization | Baseline; 3 months; 6 months; 12 months follow-up
  Self-report and military data base information regarding type, and frequency of health care received. Also, self-reports on service needs.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Schwab, PhD, Principal Investigator — The Defense and Veterans Brain Injury Center
Locations (2):
- United States (2):
  - Fort Carson, Fort Carson, Colorado
  - Fort Bragg, Fort Bragg, North Carolina

REFERENCES:
- [Derived] Ivins B, Risling M, Wisen N, Schwab K, Rostami E. Mild Traumatic Brain Injury in the Maturing Brain: An Investigation of Symptoms and Cognitive Performance in Soldiers Returning From Afghanistan and Iraq. J Head Trauma Rehabil. 2024 Jul-Aug 01;39(4):304-317. doi: 10.1097/HTR.0000000000000919. Epub 2023 Dec 7. PMID 38059837
- [Derived] Scher AI, McGinley JS, VanDam LR, Campbell AM, Chai X, Collins B, Klimp SA, Finkel AG, Schwab K, Lipton RB, Johnson KW. Plasma calcitonin gene-related peptide and nerve growth factor as headache and pain biomarkers in recently deployed soldiers with and without a recent concussion. Headache. 2023 Oct;63(9):1240-1250. doi: 10.1111/head.14635. Epub 2023 Oct 5. PMID 37796114
- [Derived] Scher AI, McGinley JS, Wirth RJ, Lipton RB, Terrio H, Brenner LA, Cole WR, Schwab K. Headache complexity (number of symptom features) differentiates post-traumatic from non-traumatic headaches. Cephalalgia. 2021 Apr;41(5):582-592. doi: 10.1177/0333102420974352. Epub 2020 Nov 27. PMID 33242991
- [Derived] Metti A, Schwab K, Finkel A, Pazdan R, Brenner L, Cole W, Terrio H, Scher AI. Posttraumatic vs nontraumatic headaches: A phenotypic analysis in a military population. Neurology. 2020 Mar 17;94(11):e1137-e1146. doi: 10.1212/WNL.0000000000008935. Epub 2020 Jan 10. PMID 31924681
- [Derived] Betthauser LM, Adams RS, Hostetter TA, Scher AI, Schwab K, Brenner LA. Characterization of lifetime TBIs in a cohort of recently deployed soldiers: The warrior strong study. Rehabil Psychol. 2019 Nov;64(4):398-406. doi: 10.1037/rep0000286. Epub 2019 Aug 1. PMID 31368742
- [Derived] Schwab K, Terrio HP, Brenner LA, Pazdan RM, McMillan HP, MacDonald M, Hinds SR 2nd, Scher AI. Epidemiology and prognosis of mild traumatic brain injury in returning soldiers: A cohort study. Neurology. 2017 Apr 18;88(16):1571-1579. doi: 10.1212/WNL.0000000000003839. Epub 2017 Mar 17. PMID 28314862